CLINICAL TRIAL: NCT00002947
Title: A Phase I Study of [111In-DTPA-D-Phe]-Octreotide in Patients With Refractory Malignancies Expressing Somatostatin Receptors
Brief Title: Indium In 111 Pentetreotide in Treating Patients With Refractory Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065414; YALE-HIC-9041; NCI-G97-1154
Record Dates: First submitted 1999-11-01; First posted 2004-03-26 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Langerhans Cell Histiocytosis; Gastrointestinal Carcinoid Tumor; Head and Neck Cancer; Intraocular Melanoma; Islet Cell Tumor; Kidney Cancer; Lung Cancer; Melanoma (Skin); Neoplastic Syndrome; Neuroendocrine Carcinoma of the Skin; Pheochromocytoma
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; gastrinoma; insulinoma; recurrent islet cell carcinoma; thyroid gland medullary carcinoma; prolactin-producing pituitary tumor; iris melanoma; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; recurrent intraocular melanoma; stage IV melanoma; recurrent melanoma; WDHA syndrome; somatostatinoma; pancreatic polypeptide tumor; glucagonoma; childhood Langerhans cell histiocytosis; metastatic pheochromocytoma; recurrent pheochromocytoma; pulmonary carcinoid tumor; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III neuroendocrine carcinoma of the skin; recurrent neuroendocrine carcinoma of the skin
MeSH Terms: conditions — Central Nervous System Neoplasms; Head and Neck Neoplasms; Uveal Melanoma; Adenoma, Islet Cell; Kidney Neoplasms; Lung Neoplasms; Melanoma; Neoplasms; Carcinoma, Merkel Cell; Pheochromocytoma; Carcinoma, Renal Cell; Small Cell Lung Carcinoma; Gastrinoma; Insulinoma; Carcinoma, Islet Cell; Carcinoma, Medullary; Vipoma; Somatostatinoma; Glucagonoma; Esthesioneuroblastoma, Olfactory | interventions — pentetreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: indium In 111 pentetreotide

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other sources to damage tumor cells. Giving radiation therapy in different ways may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of indium In 111 pentetreotide in treating patients who have refractory cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD), toxic effects, and the preliminary antitumor activity of indium In 111 pentetreotide.

OUTLINE: This is a dose escalation study. Patients receive indium In III pentetreotide (OctreoScan) IV on day 1. Imaging is conducted on days 3 and 6. Treatment continues weekly for a total of 4 courses in the absence of disease progression or unacceptable toxicity. Cohorts of at least 3 patients receive escalating doses of OctreoScan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose limiting toxicities. Patients are followed every 3 months for the first year, then every 6 months thereafter.

PROJECTED ACCRUAL: Up to 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignancy with no alternate treatments available Measurable or evaluable progressive disease Somatostatin receptors present on tumor and uptake demonstrated on diagnostic scan with OctreoScan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Platelet count at least 100,000/mm3 Absolute neutrophil count at least 1,500/mm3 Hepatic: Total bilirubin no greater than 2.0 mg/dL Renal: Creatinine clearance at least 40 mL/min Other: No active infections Not HIV positive No coexisting medical condition Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior wide field radiation therapy Surgery: Recovery from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1996-10; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Murren, MD, Study Chair — Yale University
Locations (1):
- Yale Comprehensive Cancer Center, New Haven, Connecticut, United States